CLINICAL TRIAL: NCT01025427
Title: Treating HIV-infected Elite Controllers as a Model of HIV Remission
Brief Title: HIV Persistence and Viral Reservoirs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California HIV/AIDS Research Program (Other); Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H52889-35080
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: HIV; HIV Infections
Keywords: HIV; HIV persistence; HIV reservoirs
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Elite controller (Experimental): Sixteen controllers will be treated with open-label raltegravir/tenofovir/emtricitabine for 24 weeks.
  Interventions: Drug: Raltegravir, tenofovir/emtricitabine

INTERVENTIONS:
Drug: Raltegravir, tenofovir/emtricitabine — 16 controllers will be treated with open-label raltegravir/tenofovir/emtricitabine for 24 weeks.

SUMMARY:
Although highly active antiretroviral therapy (HAART) decreases HIV-associated mortality, it does not to completely restore health. Patients doing well on otherwise effective HAART remain at risk for cancer, cardiovascular/liver disease, osteopenia, and other "non-AIDS-defining" events. While complete eradication may never be feasible, a "functional cure" in which patients are able to maintain undetectable viral loads indefinitely without therapy may be possible. The best evidence for this are the so-called "elite" controllers, whom we define as individuals who are HIV-seropositive, with plasma HIV RNA levels below the level of conventional detection without treatment. Controllers may be conceptualized as a naturally occurring model of a functional cure (or "HIV remission"), and are ideal patients in which to study HIV persistence and the possibility of eradication.

We propose to conduct a pilot study to better characterize the reservoirs that lead to viral persistence in a group of well-characterized controllers. We propose two specific aims: 1) to characterize the dynamics of viral production in blood and gut-associated lymphoid tissue (GALT) in controllers; and 2) to prospectively treat 10 controllers with raltegravir, tenofovir/emtricitabine for 24 weeks and study the effects of HAART on viral dynamics and host inflammatory responses.

Our primary hypotheses are: 1) viral replication is ongoing in untreated controllers, 2) HAART will reduce viral replication in blood and GALT and decrease immune activation, and 3) higher levels of immune activation are associated with greater measures of microbial translocation and distribution of virus to more differentiated T cell subsets.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, and
2. HIV infection, and
3. Antiretroviral-naïve, and
4. CD4+ T cell count >350 cells/mm3, and
5. "Controllers": antiretroviral untreated with 50-1000 copies/mL viral load for at least 12 months

Exclusion criteria:

1. Persons with known rheumatologic conditions (e.g., systemic lupus erythematosus), because of their predilection for biologic false-positive testing on HIV antibody tests.
2. Screening absolute neutrophil count <1,000 cells/mm3, platelet count <70,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <40 mL/minute, aspartate aminotransferase >100 units/L, alanine aminotransferase >100 units/L.
3. Screening genotype resistance testing showing resistance to tenofovir or emtricitabine.
4. Known kidney disease.
5. Known bone disease, including pathologic fractures.
6. Patients with chronic Hepatitis B infection, because of the risk of liver abnormalities after starting and stopping tenofovir/emtricitabine.
7. Concurrent treatment with lamivudine, adefovir, entecavir, or telbivudine.
8. Serious illness requiring hospitalization or parental antibiotics within the preceding 3 months.
9. Any vaccination 2 weeks prior to baseline (Day 0) visit and throughout the study period. NOTE: Because the study will most likely be actively recruiting during the influenza season, all subjects will be encouraged to receive their annual influenza vaccine at the screening visit (4 weeks prior to baseline [Day 0] visit) if they have not already been vaccinated for the 2009-10 season and if it is medically indicated.
10. Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drug in the preceding 16 weeks (e.g. corticosteroid therapy equal to or exceeding a dose of 15 mg/day of prednisone for more than 10 days, IL-2, interferon-alpha, methotrexate, cancer chemotherapy). NOTE: Use of inhaled or nasal steroid use is not exclusionary.
11. Concurrent treatment with phenobarbital, phenytoin, or rifampin.
12. Pregnant or breastfeeding women. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyu Hatano, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Hatano H, Yukl SA, Ferre AL, Graf EH, Somsouk M, Sinclair E, Abdel-Mohsen M, Liegler T, Harvill K, Hoh R, Palmer S, Bacchetti P, Hunt PW, Martin JN, McCune JM, Tracy RP, Busch MP, O'Doherty U, Shacklett BL, Wong JK, Deeks SG. Prospective antiretroviral treatment of asymptomatic, HIV-1 infected controllers. PLoS Pathog. 2013;9(10):e1003691. doi: 10.1371/journal.ppat.1003691. Epub 2013 Oct 10. PMID 24130489

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Controller
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Controller
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Estimated Ultrasensitive Plasma HIV RNA Levels Between Baseline and Week 24
Description: The isothermal transcription mediated amplification (TMA) assay (Aptima, Gen-Probe/Hologic) was used to measure ultrasensitive plasma HIV RNA levels at weeks 0, 4, 12, and 24. This is a nucleic acid-amplification test that has been FDA-approved for the early detection of HIV infection in blood donors. It is a highly specific and sensitive assay, with a singlicate 50% detection limit of 3.6-14 copies/mL. The assay was performed in triplicate on 0.5 mL plasma (1.5 mL total plasma), improving the overall 50% detection limit to < 5 copies/mL.
Time Frame: 24 weeks
Measure: Mean (95% Confidence Interval); unit: fold decrease in signal/cutoff ratio
Groups:
- HIV Controller: Sixteen asymptomatic controllers were prospectively treated with open-label raltegravir and tenofovir/emtricitabine for 24 weeks. Controllers were defined by the following inclusion criteria: (1) HIV-seropositive; (2) ART untreated; and (3) plasma HIV RNA <1,000 copies/mL for ≥12 months.
Arm/Group | HIV Controller
Number analyzed (Participants) | 16
fold decrease in signal/cutoff ratio | 66 [28 to 155]

ADVERSE EVENTS:
Arm/Group | Controller
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No